CLINICAL TRIAL: NCT06053411
Title: Pilot Study to Assess the Contribution of UGT2B17 and Associated Genetic Polymorphisms on the Pharmacokinetics of Diclofenac Alone and Upon Co-administration With Curcumin
Brief Title: Contribution of UGT2B17 to the Pharmacokinetics of Diclofenac
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Principal Investigator, Mary Paine, Professor, Washington State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20104
Record Dates: First submitted 2023-09-15; First posted 2023-09-25 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Interaction
Keywords: Pharmacokinetic
MeSH Terms: interventions — Diclofenac; Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: diclofenac alone (baseline) (Experimental): A single dose of diclofenac (25 mg capsule) will be administered by mouth to 5 participants (minimum 2 females) genotyped as extensive metabolizers (Arm 1A) and 5 participants (minimum 2 females) genotyped as poor metabolizers (Arm 1B). Plasma and urine will be collected from 0-12 hours. A washout of at least 3 days will elapse between Arm 1 and Arm 2.
  Interventions: Drug: Diclofenac
- Arm 2: diclofenac + curcumin (Experimental): A single oral dose of diclofenac (25 mg capsule) and a single oral dose of curcumin (2,000 mg tablet) will be administered by mouth to the 5 participants genotyped as extensive metabolizers. Plasma and urine will be collected from 0-12 hours.
  Interventions: Drug: Diclofenac; Dietary Supplement: curcumin

INTERVENTIONS:
Drug: Diclofenac — 25 mg capsule
  Other Names: Voltaren
Dietary Supplement: curcumin — 2,000 mg tablet
  Arms: Arm 2: diclofenac + curcumin

SUMMARY:
The purpose of this pilot study is to gather preliminary data on the (1) contribution of the understudied drug metabolizing enzyme, UDP-glucuronosyltransferase (UGT) 2B17, to the metabolism of a widely used medication, diclofenac, and (2) impact of the UGT2B17 inhibitor and natural product, curcumin, on diclofenac pharmacokinetics. Results will inform future studies aimed to assess the effects of UGT2B17 genetic polymorphisms and co-consumed xenobiotics on the pharmacokinetics and toxicity risk of diclofenac and other UGT2B17 drug substrates.

DETAILED DESCRIPTION:
Diclofenac, a widely used non-steroidal anti-inflammatory drug, has been linked to severe adverse effects such as gastrointestinal ulcers and bleeding and cardiotoxicity. Based on cardiotoxicity reports, US and European regulatory agencies withdrew over-the-counter (OTC) diclofenac, requiring the drug to be a prescription-only medication. However, diclofenac remains OTC in many countries, including Australia, China, and India, among others. Reported metabolic pathways of diclofenac in the liver are mediated by the prominent drug metabolizing enzyme, cytochrome P450 (CYP) 2C9, and the conjugative enzyme, UDP-glucuronosyltransferase (UGT) 2B7. However, recent in vitro and in silico data indicated that diclofenac is metabolized almost exclusively by a less-studied UGT, UGT2B17, in the intestine.

UGT2B17 is among the most genetically polymorphic enzymes, with highly prevalent copy number variations (CNVs). Individuals homozygous for the null allele, UGT2B17*2 (CNV=0), are considered poor metabolizers (PMs), whereas those homozygous for the reference allele, UGT2B17*1/*1 (CNV=2), are considered extensive metabolizers (EMs). Deletion of this gene may lead to large interindividual variability in the pharmacokinetics - and toxicity risk - for patients taking diclofenac and other UGT2B17 substrates, including vorinostat, MK7426, tamoxifen, exemestane, and testosterone. Collectively, considering UGT2B17 CNVs on the metabolism of these drugs is critical to ensure consistent and optimum safety, efficacy, and patient outcomes.

Recent preliminary data showed that curcumin, a principal curcuminoid of the natural product turmeric, is a potent inhibitor of UGT2B17. Turmeric is used worldwide and was the 2nd top-selling herbal supplement in the US in 2021, with nearly $100 million in total sales. Considering both turmeric/curcumin and diclofenac are used for arthritis and other inflammatory conditions, there is a high likelihood of patients co-consuming curcumin and diclofenac, raising concerns for variable diclofenac pharmacokinetics and toxicity risk.

The purpose of this pilot study is to gather preliminary data on the (1) contribution of UGT2B17 to diclofenac metabolism and (2) impact of curcumin co-administration on diclofenac pharmacokinetics. Results will inform future studies aimed to evaluate the effects of UGT2B17 genetic polymorphisms and co-consumed xenobiotics on the pharmacokinetics and toxicity risk of diclofenac and other UGT2B17 drug substrates.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18-64 years and healthy
* Not taking any medications (prescription and non-prescription) or dietary/herbal supplements known to alter the pharmacokinetics of diclofenac or curcumin
* Willing to abstain from consuming caffeinated beverages or other caffeine-containing products the evening before and morning of the first day of each study arm
* Willing to abstain from consuming any alcoholic beverages for one day prior to any study day, during the 14-hour inpatient days, and for the outpatient visit(s) following the 14-hour days
* Willing to use a secondary method of birth control that does not include the introduction or discontinuance of hormonal-based birth control (such as abstinence, copper IUD, or condoms)
* Have the time to participate
* Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for the subject to comply with the requirements of the study

Exclusion Criteria:

* Under the age of 18 or over the age of 65 years
* Smoke/vape/chew tobacco products
* Use cannabis products, including marijuana, hemp, and other THC- or CBD-containing products
* Have any current major illness or chronic illness such as (but not limited to) kidney disease, hepatic disease, diabetes mellitus, hypertension, coronary artery disease, chronic obstructive pulmonary disease, cancer, or HIV/AIDS
* History of anemia or any other significant hematologic disorder
* History of drug or alcohol addiction or major psychiatric illness
* Pregnant or nursing or plan to become pregnant within 3 weeks after participation
* History of allergy intolerance to diclofenac or curcumin
* Taking concomitant medications, both prescription and non-prescription (including dietary supplements/herbal products), known to alter the pharmacokinetics of diclofenac or curcumin
* Taking any turmeric spice or curcumin supplement
* Presence of a condition or abnormality that, in the opinion of the Investigator, would compromise participant safety or quality of the data
* Out-of-range clinical laboratory value that the study physician considers participation in the study a health risk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-18 (Estimated); Study Completion 2026-08-18 (Estimated)

PRIMARY OUTCOMES:
Diclofenac area under the concentration vs. time curve (AUC) in UGT2B17 extensive metabolizers (EMs) | 0-12 hours
  Diclofenac AUC in UGT2B17 EMs
Diclofenac AUC in poor metabolizers (PMs) | 0-12 hours
  Diclofenac AUC in UGT2B17 PMs
Diclofenac AUC in EMs in the presence of curcumin | 0-12 hours
  Diclofenac AUC in UGT2B17 EMs in the presence of curcumin
Diclofenac maximum concentration (Cmax) in EMs | 0-12 hours
  Diclofenac Cmax in UGT2B17 EMs
Diclofenac Cmax in PMs | 0-12 hours
  Diclofenac Cmax in UGT2B17 PMs
Diclofenac Cmax in EMs in the presence of curcumin | 0-12 hours
  Diclofenac Cmax in UGT2B17 EMs in the presence of curcumin
Diclofenac renal clearance (CLr) in EMs | 0-12 hours
  Diclofenac CLr in UGT2B17 EMs
Diclofenac CLr in PMs | 0-12 hours
  Diclofenac CLr in UGT2B17 PMs
Diclofenac CLr in EMs in the presence of curcumin | 0-12 hours
  Diclofenac CLr in UGT2B17 EMs in the presence of curcumin
Diclofenac half-life (t1/2) in EMs | 0-12 hours
  Diclofenac t1/2 in UGT2B17 EMs
Diclofenac half-life (t1/2) in PMs | 0-12 hours
  Diclofenac t1/2 in UGT2B17 PMs
Diclofenac half-life (t1/2) in EMs in the presence of curcumin | 0-12 hours
  Diclofenac t1/2 in UGT2B17 EMs in the presence of curcumin

CONTACTS AND LOCATIONS:
Locations (1):
- Washington State University College of Pharmacy and Pharmaceutical Sciences, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schjerning AM, McGettigan P, Gislason G. Cardiovascular effects and safety of (non-aspirin) NSAIDs. Nat Rev Cardiol. 2020 Sep;17(9):574-584. doi: 10.1038/s41569-020-0366-z. Epub 2020 Apr 22. PMID 32322101
- [Background] Whirl-Carrillo M, Huddart R, Gong L, Sangkuhl K, Thorn CF, Whaley R, Klein TE. An Evidence-Based Framework for Evaluating Pharmacogenomics Knowledge for Personalized Medicine. Clin Pharmacol Ther. 2021 Sep;110(3):563-572. doi: 10.1002/cpt.2350. Epub 2021 Jul 22. PMID 34216021
- [Background] Ahire D, Heyward S, Prasad B. Intestinal Metabolism of Diclofenac by Polymorphic UGT2B17 Correlates with its Highly Variable Pharmacokinetics and Safety across Populations. Clin Pharmacol Ther. 2023 Jul;114(1):161-172. doi: 10.1002/cpt.2907. Epub 2023 Apr 29. PMID 37042794
- [Background] Xue Y, Sun D, Daly A, Yang F, Zhou X, Zhao M, Huang N, Zerjal T, Lee C, Carter NP, Hurles ME, Tyler-Smith C. Adaptive evolution of UGT2B17 copy-number variation. Am J Hum Genet. 2008 Sep;83(3):337-46. doi: 10.1016/j.ajhg.2008.08.004. Epub 2008 Aug 28. PMID 18760392
- [Background] Wang YH, Trucksis M, McElwee JJ, Wong PH, Maciolek C, Thompson CD, Prueksaritanont T, Garrett GC, Declercq R, Vets E, Willson KJ, Smith RC, Klappenbach JA, Opiteck GJ, Tsou JA, Gibson C, Laethem T, Panorchan P, Iwamoto M, Shaw PM, Wagner JA, Harrelson JC. UGT2B17 genetic polymorphisms dramatically affect the pharmacokinetics of MK-7246 in healthy subjects in a first-in-human study. Clin Pharmacol Ther. 2012 Jul;92(1):96-102. doi: 10.1038/clpt.2012.20. Epub 2012 Jun 6. PMID 22669291